CLINICAL TRIAL: NCT06150846
Title: Sperm Video Recording Protocol
Status: Active, not recruiting | Type: Observational
Sponsor: BAIBYS Fertility (Industry)
Responsible Party: Sponsor
Other Study IDs: BCP-002 Sperm VR Trial
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Sperm Classification
Keywords: Sperm; Artificial Inteligence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to obtain anonymous video clips of male semen at high magnification, to manually select out of the video spermatozoon images, and to manually classify their morphology by qualified embryologists based on the WHO Manual criteria in order to train the BAIBYS™ Fertility System. The study will enroll males attending the clinic who may elect to contribute their unused excess sample materials from semen analysis or IVF/ICSI (Intracytoplasmic sperm injection) which is a technique used during in vitro fertilization (IVF).

DETAILED DESCRIPTION:
The study will obtain video clips of 40 male subjects semen sample at high magnification. Each subject contributes 1 sample from which 10 minutes of video is recorded.

A total of 720,000 frames are expected to be collected at 30 frames per second. At least 6,000 frames will be selected at random from these 10,800-14,500 frames to be labeled by at least two embryologists. The sperm morphology will be rated according to the Kruger criteria per the WHO 6th edition. The data collected will be utilized to train the Artificial Intelligence (AI) used within the BAIBYS System.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth and possessing typical male anatomy (i.e., one or two testicles and penis)
* Scheduled to produce a semen sample for fertility evaluation
* Able to produce a semen sample, including, in the judgement of the PI, ability to follow instructions provided in English by the physician or physician's team members
* At least a 10th grade education level, to be able to read and understand the ICF; evaluated by either completion of 10th grade, or by any higher level of education or GED
* Age 22 or older at the time of consent

Exclusion Criteria:

* Known azoospermia prior to semen analysis.
* Subjects with azoospermia or otherwise inadequate sample discovered during the trial will be compensated for their participation in recognition of their efforts to contribute to science, but will be replaced with an additional subject for the data collection and labeling to reach a total sample of up to 40 videos
* History of chemotherapy or radiation within prior 12 months, due to increased chance of azoospermia
* Developmental delays or other neurological impairment that could impair ability to freely consent, as evaluated by the PI
* Any reason why in the sole judgement of the PI, consent to participate cannot be freely given

Min Age: 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male at birth and possessing typical male anatomy (i.e., one or two testicles and penis)
Study Population: The study will enroll 30-40 male subjects attending the clinic and willing to contribute their unused excess sample materials from semen analysis or IVF/ICSI. Enrollment will include three sub-populations of at least 15 patients to ensure diversity [characteristics of ethnic and racial diversity, BMI diversity, and normal (> WHO 5%ile cutoffs) versus abnormal morphology].
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Obtaining 6,000 classified sperm images | Each semen sample will be recorded for 10 minutes
  Obtaining 6,000 sperm images classified each by at least 2 embryologist based on the WHO 6th edition criteria to add to the AI training of the Baibys system.

CONTACTS AND LOCATIONS:
Overall Officials: Carter Owen, M.D., Principal Investigator — CCRM Fertility Clinic and IVF Clinic
Locations (1):
- CCRM Northern Virginia, Vienna, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient's data including selection of sperm images/videos will be used together with the clinical study report and protocol will be shared to the medical writer and the supervisor author for the purpose of the the final publication.
Supporting Information: Study Protocol, CSR
Time Frame: 12 months after follow up pivotal trial is completed
Access Criteria: The IPD will be anonymized and shared as described in the plan. All those getting access will not be able to de-identify any patient's data.
  Anonymized patient's data including selection of sperm images/videos will be used together with the clinical study report and protocol will be shared to the medical writer and the supervisor author for the purpose of the the final publication.